CLINICAL TRIAL: NCT02812173
Title: Prospective, Randomized, Three-arm, Open Controlled Trial Comparing the Quality of Micturition and the Patient Comfort by Various Urinary Drainage After Robot-assisted Radical Prostatectomy (RARP)
Brief Title: Postoperative Patient Comfort and Quality of Micturition in Suprapubic Tube vs. Transurethral Catheterization After RARP
Acronym: MPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital Gronau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: U4DGYZXT2DBN
Record Dates: First submitted 2016-05-18; First posted 2016-06-24 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
Keywords: urinary drainage; urethral catheter; suprapubic tube; pain; discomfort; radical prostatectomy; robotic surgery; urinary infection
MeSH Terms: conditions — Prostatic Neoplasms; Pain; Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- suprapubic tube ex 2 day (Active Comparator): patients who underwent robot-assisted radical prostatectomy and got intraoperatively, a suprapubic tube, which was withdrawn on the 2th day after the surgery
  Interventions: Device: suprapubic tube ex 2 day
- suprapubic tube ex 5 day (Active Comparator): patients who underwent robot-assisted radical prostatectomy and got intraoperatively, a suprapubic tube, which was withdrawn on the 5th day after the surgery
  Interventions: Device: suprapubic tube ex 5 day
- transurethral catheter ex 5 day (Active Comparator): patients who underwent robot-assisted radical prostatectomy and got intraoperatively, a transurethral catheter, which was withdrawn on the 5th day after the surgery
  Interventions: Device: transurethral catheter ex 5 day

INTERVENTIONS:
Device: suprapubic tube ex 2 day — balloon catheter for suprapubic bladder-drainage, suprapubic tube removal on the second day after the surgery
  Other Names: Uromed
  Arms: suprapubic tube ex 2 day
Device: suprapubic tube ex 5 day — balloon catheter for suprapubic bladder-drainage, suprapubic tube removal on the fifth day after the surgery
  Other Names: Uromed
  Arms: suprapubic tube ex 5 day
Device: transurethral catheter ex 5 day — transurethral catheter withdrawal removal on the fifth day after the surgery
  Other Names: Uromed
  Arms: transurethral catheter ex 5 day

SUMMARY:
The purpose of the study is to determine, whether the postoperative quality of micturition and continence can be improved depending on the urinary drainage catheter and retention after robot assisted radical prostatectomy. Another finding could be the study of the pain assessment of the patient, as well as the pain medication at the various derivatives. Further check whether infections and the presence of bacteriuria can be reduced or avoided by the form of urinary drainage.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 Years
* Voluntarily agreement to participate in this study
* filled in and signed Informed Consent
* release of medical records for regulatory or research purposes
* clinically organ-confined prostate cancer
* recommended and planned robot-assisted radical prostatectomy

Exclusion Criteria:

* Participation in other interventional trials that could interfere with the present study
* International Prostate Symptom Score (IPPS) > 18
* History of radiation or chemotherapy
* History of transurethral prostate resection
* unable to provide informed consent
* unwillingness to storage and forwarding of pseudonymous data

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Urinary leakage measured by pad test in grams | within the day 2 or day 5 after the surgery for 24 hours

SECONDARY OUTCOMES:
Detection of postoperative pain related to urinary drainage by numeric rating scale (NRS) | once a day, first 7 days after the surgery
Recording of complications | within the 4 weeks after surgery
Urine status measured by flow cytometry | within the day 2 or day 5 after the surgery
Residual urine measured by bladder scan in ml | 3 times within the day 2 or day 5 after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nina Harke, MD., Principal Investigator — St. Antonius Hospital Gronau; Mustapha Addali, MD., Study Chair — St. Antonius Hospital Gronau
Locations (1):
- Department of Urology, Pediatric Urology and Urologic Oncology, St. Antonius Hospital Gronau, Gronau, Germany

IPD SHARING:
Plan to Share IPD: No